CLINICAL TRIAL: NCT02132585
Title: Cross Sectional Study of Use of Speckle Tracking Echocardiography in the Early Diagnosis of Cardiovascular Dysfunction and Performance in Sjogren Patients
Brief Title: Cross-sectional Study of Use of Speckle Method in Early Diagnosis of Cardiovascular Dysfunction
Acronym: SPEEDCARS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianturco Luigi, MD, University of Roma La Sapienza
Other Study IDs: Spk-001
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-02

CONDITIONS: Sjogren Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sjogren: Sjogren Patients evaluated with Speckle tracking echocardiography
  Interventions: Procedure: Speckle tracking echocardiography
- Control: Controls Speckle tracking echocardiography
  Interventions: Procedure: Speckle tracking echocardiography

INTERVENTIONS:
Procedure: Speckle tracking echocardiography

SUMMARY:
Speckle tracking (STE) is a novel echocardiographic technique which permits calculation of myocardial velocities and deformation parameters such as strain and strain rate (SR). It is demonstrated that these parameters provide important insights into systolic and diastolic function, ischaemia, myocardial mechanics and many other pathophysiological processes of the heart. In this preliminary study, we investigated the role of STE in detection of early ventricular dysfunction in patients with Sjogren Syndrome, focusing on cardiorespiratory fitness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Sjogren Syndrome

Exclusion Criteria:

* previous cardiovascular events
* unstable angina
* stroke
* diagnosis of heart failure
* incapacity to provide an informed consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients enrolled from cardiovascular clinic
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Myocardial Strain reduction in Sjogren Patients | Baseline, 24 weeks
  Longitudinal Myocardial Strain reduction could be an early marker of cardiac dysfunction in patients with Sjogren Syndrome, significantly better than common measurement (such as ejection fraction)

SECONDARY OUTCOMES:
Association between 6minute-walking-test and Longitudinal strain reduction | baseline, 24 weeks
  Longitudinal strain reduction could be linked to decrease in cardiorespiratory fitness, especially in 6-minute-walking-test

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Galeazzi IRCCS of Milan, Milan, Italy
  - Sapienza University, Rome